CLINICAL TRIAL: NCT03686722
Title: Effect of Co-administration of Metformin and Daclatasvir on the Pharmacokinetics and Pharmacodynamics of Metformin
Brief Title: Effect of Co-administration of Metformin and Daclatasvir on the Pharmacokinetis and Pharmacodynamics of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohamed Raslan (Other)
Collaborators: Ain Shams University (Other); Drug Research Centre, Cairo, Egypt (Other)
Responsible Party: Sponsor-Investigator, Mohamed Raslan, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MET-DAC\DDIS\01217
Record Dates: First submitted 2018-09-23; First posted 2018-09-27 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2; Hepatitis C; Drug Interactions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hepatitis C | interventions — Metformin; daclatasvir

STUDY DESIGN:
Intervention Model Description: Twenty Eligible Adult Subjects Will be Randomized Equally into two Groups: A and B To Receive Either:
  Group (A):10 subjects will receive 500 mg Metformin twice daily on day 1-4 then 1000mg metformin twice on day 5-7 Group (B):10 subjects will receive 500 mg co-administered daily with Daclatasvir 60 mg once daily on day 1-4 then 1000mg Metformin co-administered twice daily with Daclatasvir 60 mg once daily on day 5-7
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Subjects administered Metformin 500mg(Glucophage tablets) twice daily till day(4) then Metformin 1000mg twice daily till day(7)
  Interventions: Drug: Metformin
- Metformin and Daclatasvir (Experimental): Subjects Coadministered Metformin 500mg(Glucophage tablets) twice daily and Daclatasvir 60mg tablets once daily till day (4) then Metformin 1000mg twice daily and Daclatasvir 60mg tablets once daily till Day(7)
  Interventions: Drug: Metformin; Drug: Daclatasvir

INTERVENTIONS:
Drug: Metformin — Metformin is used primarly in treatment of diabetes type II
Drug: Daclatasvir — Daclatsvir is a direct acting antiviral drug
  Arms: Metformin and Daclatasvir

SUMMARY:
A Randomized,Two-period, Crossover Study to Determine the Possibility of Drug-drug Interaction After Co-administration of Metformin and Daclatasvir Where Twenty Eligible Adult Subjects Will be Randomized to Receive Either Metformin Only and/or Metformin Co-administered With Daclatasvir to measure primary outcomes including pharmacokinetics parameters as: Maximum drug concentration in plasma(Cmax), Area under the Plasma concentration Versus Time Curve from time 0 to 12 hours(AUC0-12), Clearance(CL)

DETAILED DESCRIPTION:
Study Design:

A randomized, one-way, single blinded, two-period, crossover study in adult human healthy egyptian volunteers

Methodology:

period (I): Group A:10 volunteers will receive 500 mg Metformin twice daily on day 1-4 then 1000mg metformin twice on day 5-7

GroupB:10 volunteers will receive 500 mg Metformin twice daily + Daclatasvir (DCV) 60 mg once daily on day 1-4 then 1000mg metformin twice daily+DCV 60 mg once daily on day 5-7

period (II): Group A:10 volunteers will receive 500 mg Metformin twice daily + Daclatasvir (DCV) 60 mg once daily on day 1-4 then 1000mg metformin twice daily+DCV 60 mg once daily on day 5-7

Group B:10 volunteers will receive 500 mg Metformin twice daily on day 1-4 then 1000mg metformin twice daily on day 5-7

All drug administration will be followed by 240 ml of water after at least 10 hours fasting prior to administration.

The two treatment periods will be separated by a one week washout period

Blood Sampling will be collected at a pre-dosing and at 0.25, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12 hours Urine samples will be collected for metformin analysis from 0 to 12 hours after drug administration.

A 75 g Oral glucose tolerance test(OGTT) will be carried out by ingestion of 75g glucose in 240ml water 2-hours post dosing and blood samples for determining glucose concentration during OGTTs were collected immediately before and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, and 3 hours after glucose ingestion.

Blood samples will be collected from each volunteer prior to drug administration (blank) at the predetermined sampling intervals after drug administration in ethylene diamine tetra-acetic acid(kEDTA) containing tubes.

These samples will be centrifuged and the plasma harvested and stored at -80°C until assay.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18-55 years at screening.
2. Subject has a Body Mass Index of 18 to 35 kg/m2.
3. Subject are non smokers or moderate smokers(not more than 10 cigarettes per day)
4. Subjects is willing to participate and give their final written consent prior to the commencement of the study procedures
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, and results of biochemistry, hematology and urine analysis testing within 4 weeks prior to study.
6. Subject has a normal blood pressure and pulse rate, according to the reference normal ranges.

Exclusion Criteria:

1. Treatment with any known enzyme-inducing/inhibiting agents prior to the start of the study and throughout the study.
2. Subjects who have taken any medication two weeks preceding of the trial starting date.
3. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
4. Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
5. Gastrointestinal diseases.
6. Renal diseases.
7. Cardiovascular diseases specially transient ischemic attacks and cardiac dysrhythmia .
8. Pancreatic disease including diabetes.
9. Hepatic diseases as hepatic failure, cirrhosis, galactose intolerance, fructose intolerance, glycogen storage diseases
10. Hematological disease or pulmonary disease
11. Abnormal laboratory values.
12. Subjects who have donated blood or who have been involved in a drug study within 6 weeks preceding the start of the study.
13. Positive HIV test.
14. History of or current abuse of drugs, alcohol or solvents.
15. Endocrine disorders as Pheochromocytoma, Addison disease, glucagon deficiency, carcinomas, extrahepatic tumors
16. Autoimmune disorders as Graves disease
17. Central nervous system (CNS) disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
(AUC0→12) | From first sampling interval(time zero) up to 12 hours
  Area under the plasma concentration-time curve measured in (nanogram(ng).hr/ml)
Area under the plasma concentration-time curve from time 0 to infinity (AUC0→∞) | From first sampling interval up to infinity
  Area under the plasma concentration-time curve from time 0 to infinity measured in(ng.hr/ml)
Area under the plasma concentration-time curve from time 0 to tau(AUC0→tau) | From first sampling interval up to dosing interval(Tau)
  Area under the plasma concentration-time curve from time 0 to tau measured in(ng.hr/ml)
Maximum drug concentration in plasma at steady state(Cpss) | Time corresponding to maximum drug concentration in plasma at steady state
  Maximum drug concentration in plasma at steady state measured in (ng/ml)
Half life( t½) of drug in plasma | Up to 12 hours
  Half life of drug measured in Hours(hr)
Mean residence time of drug(MRT) | From first sampling interval up to 12 hours
  Mean residence time of drug in plasma measured in (hr)
steady state Clearance of drug(CLss) | From first sampling interval up to 12 hours
  steady state Clearance of drug measured in (ml/min)
Renal Clearance of drug(CLr) | From first sampling interval up to 12 hours
  Renal Clearance of drug measured in (ml/min)
Cumulative amount of drug eliminated in urine (Ae) | From first sampling interval up to 12 hours
  Cumulative amount of drug eliminated in urine measured in (microgram(ug)/ml)
Maximum excretion rate (Urate max) | From first sampling interval up to 12 hours
  Maximum excretion rate for the drug measured in (milligram(mg)/hr)

SECONDARY OUTCOMES:
Blood Glucose(BG) levels | up to 3 hours
  Blood glucose levels measured in (mg/dl)
Area under the BG-time curve(AUG)0-3hr | up to 3 hours
  Area under the BG-time curve measured in (mg.hr/dl)
Maximum Glucose concentration(Gmax) | up to 3 hours
  Maximum Glucose concentration measured in (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Raslan, Principal Investigator — Ainshams university
Locations (1):
- Drug research centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No